CLINICAL TRIAL: NCT03679429
Title: NBI Versus White Light Endoscopy for Optical Characterization of Neoplastic Polyps in the Colorectum - the ADOPTION II Study
Brief Title: NBI Versus White Light Endoscopy for Optical Characterization of Neoplastic Polyps in the Colorectum
Acronym: ADOPTION II
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Peter Klare, Dr. med. Peter Klare, Technical University of Munich
Other Study IDs: ADOPTION II
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Colon Adenoma; Colorectal Carcinoma; Hyperplastic Polyp; Serrated Adenoma
Keywords: Colonoscopy; Adenoma detection rate; Narrow band imaging; Optical biopsy; Accuracy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colon polyps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients from the control group will be examined using a CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope. If colon polyps are detected optical diagnosis will be determined WITHOUT using the NBI function of the scope.
- Intervention: Patients from the control group will be examined using a CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope. If colon polyps are detected optical diagnosis will be determined by using the NBI function of the scope.
  Interventions: Device: NBI Function

INTERVENTIONS:
Device: NBI Function — In the intervention arm polyps will be optically characterized using the NBI function. The WASP (Workgroup serrAted polypS and Polyposis) classification will be used in order to determine the optical diagnosis.
  Other Names: NBI Function integrated in the CF-HQ 190 EVIS Exera III Advanced Diagnostic Video Colonoscope
  Groups: Intervention

SUMMARY:
Adenomas, serrated adenomas and hyperplastic polyps are polypoid lesion in the colorectum. At the present moment, all polyps should be resected endoscopically, although only adenomas and serrated adenomas, but not hyperplastic polyps have the potential to develop colorectal cancer. This approach enables the conduction of microscopic investigations of the lesions. By today, only the pathological diagnosis can distinguish exactly between these three polyp entities. Some studies have investigated the value of the optical characterization approach which is based on visual assessment of the polyp' surface structures. Based upon optical polyp features users are encouraged to predict histopathological polyp diagnoses solely on behalf of optical or endoscopical criteria. This method is conducted in real time during colonoscopy. If it could be shown, that endoscopist using the optical characterization approach are able to predict histopathological diagnoses of colonic polyps sufficiently this would possibly lead to simplification of diagnostic procedures. For instance, it would be conceivable to resect small polyps and discard them without further assessment by a pathologist. One problem in this context is a correct differentiation between hyperplastic polyps and serrated adenomas. These two polyp entities are known to show similar optical features. However, while serrated adenomas are premalignant lesions hyperplastic polyps have benign histology and never develop into cancer. It is therefore important to sufficiently distinguish hyperplastic polyps from serrated lesions.

In this study we want to investigate whether the use of narrow-band imaging (NBI) would be capable to rise accuracy of optical polyp predictions compared to standard HD white light endoscopy. NBI is a light filter tool which can be activated by pressing a button at the endoscope. The use of NBI leads to an endoscopic picture which appears blue and enables endoscopists to better assess surface structures and vascular patterns.

In a prospective randomised multicenter setting we plan to conduct colonoscopy in 370 patients. Half of the patients will be examined without the use of NBI (control arm). In these cases colonoscopists will assess optical diagnosis of polyps without turning on the NBI tool. If polyps are detected in patients belonging to the intervention arm NBI will be used and optical diagnosis will be determined using the WASP (Workgroup serrAted polypS and Polyposis) classification. All polyps will be resected and send to pathology for further microscopic assessment. After completing the trial we aim to compare accuracy of the optical diagnosis in both groups. Our hypothesis is, that by using NBI accordance between optical and histopathological diagnosis can be increased from 80% to 90%.

ELIGIBILITY:
Inclusion Criteria:

* medical indication for colonoscopy
* age ≥ 40 years
* written consent given by patient

Exclusion Criteria:

* age < 40 years
* patients denying written consent
* pregnant women
* ASA class IV, V and VI
* known contraindication for polyp resection
* indication for colonoscopy: preknown adenoma/polyp/carcinoma or inflammatory bowel disease
* indication for colonoscopy: emergency (e.g. severe rectal bleeding)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the three participating study centers (Munich, Erlangen, Stuttgart). Two of the three centers are tertiary referral-centres whereas the last one is a major regional hospital. All patients undergo colonoscopy for medical indications.
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy optical biopsy | up to 2 weeks (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks)
  After obtaining the histopathological diagnosis of resected polyps (approximately 3 days - 2 weeks after colonoscopy ) accuracy of optical diagnosis can be determined

SECONDARY OUTCOMES:
Adenoma detection rate | up to 2 weeks (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — Klinikum rechts der Isar der Technischen Universität München; Roland M Schmid, Professor, Study Director — Klinikum rechts der Isar der Technischen Universität München; Timo Rath, Professor, Study Chair — Universitätsklinikum Erlangen; Jan Peveling-Oberhag, MD, Study Chair — Robert Bosch-Krankenhaus Stuttgart
Locations (3):
- Germany (3):
  - Klinik für Innere Medizin II am Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria
  - Universitätsklinikum Erlangen, Medizinische Klinik 1, Erlangen
  - Robert-Bosch-Krankenhaus, Stuttgart

IPD SHARING:
Plan to Share IPD: No